CLINICAL TRIAL: NCT00885573
Title: Measurement of Pharyngeal Sensitivity With the SENSITEST Device: Validation of the Diagnosis Algorithm for Sleep Disordered Breathing
Brief Title: Pharyngeal Sensitivity in Diagnosis Algorithm for Sleep Apnea Syndrome
Acronym: SENSITEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: University of Liege (Other); Poitiers University Hospital (Other); University Hospital, Geneva (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 0808; 2008-A00451-54 (Registry Identifier: ID RCB)
Record Dates: First submitted 2009-04-21; First posted 2009-04-22 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-05

CONDITIONS: Sleep Apnea Syndrome
Keywords: sleep apnea; pharyngeal sensitivity; pharyngeal dilator reflex; diagnosis algorithm; patients with suspected sleep apnea syndrome
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sleep apnea subjects (Other): Patients with suspected sleep apnea syndrome will have nocturnal polysomnography. According to the number of respiratory events per hour of sleep, patients will be classified as "sleep apnea" or "controls". All the patients will be blindly assessed for pharyngeal sensitivity the morning following the nocturnal recording.
  Interventions: Device: Measurement of pharyngeal sensitivity (SENSITEST)

INTERVENTIONS:
Device: Measurement of pharyngeal sensitivity (SENSITEST) — Measurement of pharyngeal sensitivity using the SENSITEST the morning following the nocturnal polysomnographic recording to diagnose sleep disordered breathing.

SUMMARY:
Pharyngeal sensitivity is a determinant parameter of pharyngeal functioning, particularly regarding protective dilator reflexes of upper airway. Preliminary results have suggested that the use of this parameter in diagnosis algorithm such as linear discriminant analysis and random forest could predict the presence of sleep apnea syndrome in almost 98% of patients. Our study aims at validating a new diagnosis method of sleep disordered breathing which will be compared with nocturnal polysomnography, the reference method to diagnose sleep disordered breathing. Pharyngeal sensitivity will be measured using the SENSITEST device which allows an automatic measurement of the pharyngeal sensation. The use of this parameter in diagnosis algorithm will be compared with polysomnographic results.

ELIGIBILITY:
Inclusion Criteria:

* consecutively included patients with suspicion of sleep apnea syndrome
* patients who have signed the informed consent form
* patients with body mass index less than or equal 30 kg/m2

Exclusion Criteria:

* body mass index more than 30 kg/m2
* pharyngeal infection or allergic rhinitis less than 2 weeks before recordings
* craniofacial anomalies and/or limited mouth opening and/or teeth position compromising mouthpiece installation and stability during measurement
* instable dentures
* exaggerated gag reflex preventing pharynx examination
* no visibility of the soft palate
* systemic or topical anti-inflammatory treatments
* treatments that may increase the occurence of nocturnal respiratory events and/or leading to daytime sleepiness and cognitive impairment
* cardiac failure, or symptoms suggesting cardiac failure
* history of stroke
* contraindication for using xylocaine spray
* no affiliation to national insurance
* patient participating in another research study involving drugs that may interfere with sleep recordings and/or measurement of pharyngeal sensation
* patient subjected to exclusion period following participation in another research study

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2008-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
We aim to compare the novel diagnosis method with nocturnal polysomnography which is the reference method to diagnose sleep disordered breathing. | Measurement performed the morning following the nocturnal polysomnography

SECONDARY OUTCOMES:
We will determine the severity of sleep apnea for which pharyngeal sensitivity is predictive of sleep apnea syndrome. To simplify the procedure, we will precise the role of pharyngeal anesthesia in the diagnostic predictive value of the algorithm. | similar to primary outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: Maurice DEMATTEIS, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (5):
- France (4):
  - Annemasse-Bonneville Hospital, Annemasse
  - University Hospital of Grenoble, Grenoble
  - Clinic of Louvière, Lille
  - Poitiers University Hospital, Poitiers
- University Hospital of Geneva, Geneva, Switzerland

REFERENCES:
- [Background] Dematteis M, Levy P, Pepin JL. A simple procedure for measuring pharyngeal sensitivity: a contribution to the diagnosis of sleep apnoea. Thorax. 2005 May;60(5):418-26. doi: 10.1136/thx.2003.015032. PMID 15860719
- [Background] Larsson H, Carlsson-Nordlander B, Lindblad LE, Norbeck O, Svanborg E. Temperature thresholds in the oropharynx of patients with obstructive sleep apnea syndrome. Am Rev Respir Dis. 1992 Nov;146(5 Pt 1):1246-9. doi: 10.1164/ajrccm/146.5_Pt_1.1246. PMID 1443879
- [Background] Kimoff RJ, Sforza E, Champagne V, Ofiara L, Gendron D. Upper airway sensation in snoring and obstructive sleep apnea. Am J Respir Crit Care Med. 2001 Jul 15;164(2):250-5. doi: 10.1164/ajrccm.164.2.2010012. PMID 11463596
- [Background] Guilleminault C, Li K, Chen NH, Poyares D. Two-point palatal discrimination in patients with upper airway resistance syndrome, obstructive sleep apnea syndrome, and normal control subjects. Chest. 2002 Sep;122(3):866-70. doi: 10.1378/chest.122.3.866. PMID 12226025
- [Background] Woodson BT, Garancis JC, Toohill RJ. Histopathologic changes in snoring and obstructive sleep apnea syndrome. Laryngoscope. 1991 Dec;101(12 Pt 1):1318-22. doi: 10.1002/lary.5541011211. PMID 1766303
- [Background] Friberg D. Heavy snorer's disease: a progressive local neuropathy. Acta Otolaryngol. 1999;119(8):925-33. doi: 10.1080/00016489950180306. PMID 10728936
- [Background] Boyd JH, Petrof BJ, Hamid Q, Fraser R, Kimoff RJ. Upper airway muscle inflammation and denervation changes in obstructive sleep apnea. Am J Respir Crit Care Med. 2004 Sep 1;170(5):541-6. doi: 10.1164/rccm.200308-1100OC. Epub 2004 May 19. PMID 15151922
- [Background] Mayer P, Dematteis M, Pepin JL, Wuyam B, Veale D, Vila A, Levy P. Peripheral neuropathy in sleep apnea. A tissue marker of the severity of nocturnal desaturation. Am J Respir Crit Care Med. 1999 Jan;159(1):213-9. doi: 10.1164/ajrccm.159.1.9709051. PMID 9872841
- [Background] Deegan PC, McNicholas WT. Pathophysiology of obstructive sleep apnoea. Eur Respir J. 1995 Jul;8(7):1161-78. doi: 10.1183/09031936.95.08071161. PMID 7589402
- [Background] Young T, Palta M, Dempsey J, Skatrud J, Weber S, Badr S. The occurrence of sleep-disordered breathing among middle-aged adults. N Engl J Med. 1993 Apr 29;328(17):1230-5. doi: 10.1056/NEJM199304293281704. PMID 8464434